CLINICAL TRIAL: NCT04779398
Title: Investigating Associations Between Chronic Electronic Device Blue Light Exposure, Dietary Xanthophyll Intake and Macular Pigment Density in Humans.
Brief Title: Association of MPOD Values With Blue Light.
Acronym: AMPBL19
Status: Completed | Type: Observational
Sponsor: The University of Queensland (Other)
Responsible Party: Sponsor
Other Study IDs: 2019002736
Record Dates: First submitted 2021-01-24; First posted 2021-03-03 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Age Related Macular Degeneration
Keywords: macular pigment optical density; lutein; zeaxanthin; dietary intake; blue light
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma blood sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to investigate in healthy adults 18-65 years of age the association of electronic device blue light exposure and macular pigment optical density (MPOD) considering usual dietary intake of lutein and zeaxanthin (L/Z) as confirmed by serum lutein and zeaxanthin concentrations.

It is hypothesised in healthy adults 18-65 years of age:

1. Higher usual daily electronic device blue light exposure will be negatively correlated with MPOD value.
2. Usual dietary intake of L/Z will be positively correlated with MPOD value.
3. L/Z concentration will be positively correlated with MPOD value.
4. Usual dietary intake of L/Z will be positively correlated with plasma L/Z concentrations.
5. Higher usual intake of L/Z will mitigate the effect of higher electronic device exposure on MPOD value.

DETAILED DESCRIPTION:
Exponential uptake of modern technology over the last 30 years (computers) and 10 years (smartphones) has resulted in remarkable increase in artificial blue light exposure amongst all age groups. This suggests the incidence of age-related macular degeneration (AMD) could be increasing significantly in the population in the years to come. It is unknown whether the extent of daily blue light exposure influences macular pigment optical density (MPOD) in young to middle age adults. Stringham et al. (2017) showed that, in 18-25 year old healthy adults, exposed to electronic devices over 6 hours daily, MPOD value and visual performance significantly improved after 6 months of lutein/zeaxanthin/meso-zeaxanthin supplementation. The findings of this project may inform on the risks of high exposure to electronic screens and the need to address with preventive measures the potential decline in MPOD and increased risk of AMD. The impact of usual dietary intake of macular xanthophylls on circulating concentrations and MPOD will be investigated. Findings may inform guidelines on recommended daily intake of these food constituents either through diet or supplementation.

Data Management and Confidentiality of Data Collected:

Consent is sought for extended use of the collected data which means it may be used in future research. For example, in the future if more sensitive methods for detecting L/Z, or other macular pigments become available, stored blood samples may be re-analysed. Furthermore, data may be used for subsequent statistical analysis and statistical analysis may be published in peer-reviewed journals, however no identifiable personal details will be published or used. Any personal information, such as full name and date of birth will remain confidential to only the study investigators at all times.

All hard copy personal information and measures taken as part of the study protocol will be stored in locked filing cabinets when not in use, and will only be accessible to approved study investigators. Any electronic data collected for the study will be stored using the UQ Research Data Management system. Data will be de-identified through the use of participant ID numbers allocated at enrolment. Re-identification of participant information will only be accessible by study investigators. At the conclusion of the study, participant hard copy files and trial documents are kept in locked filing cabinets for a period of 15 years. After this time, records will be disposed of by a certified record destruction, such as shredding.

Blood samples will be collected for research purposes, specifically for the measurement of plasma lutein and zeaxanthin concentrations. Collected samples will be stored as per the extended consent sought, held for up to 15 years. After this time, they will be destroyed via incineration. Collected plasma samples will only be identifiable via the participant study number allocated at enrolment. All publicly shared data or data used in publications will be in a non-identifiable form.

Data recorded and maintained for this trial will be controlled in accordance with the national Privacy Principles and Privacy Act 1988.

Sample Size:

Sample size calculation was performed on the basis of a MPOD coefficient of variation of 0.187 optical density units (ODU) measured in a sample of 5581 adults using the Macular Pigment Screener II (18). A minimum of 105 participants was calculated using a two tailed, random model, linear multiple regression with an alpha error probability: 0.05, power: 0.90, number of predictors: 4. This also allows for a 20% drop out rate.

Statistical Tests:

Analysis will be conducted using GraphPad Prism 8. Participants will be stratified by MPOD.

1. Descriptive statistics will be performed.
2. All data will be tested for normality of distribution using the D'Agostino-Pearson normality test.
3. Based on the outcome of testing for normality of distribution, Spearman or Pearson's correlations will be used to test for correlation between the following variables.

   1. MPOD and daily hours of electronic device use.
   2. MPOD and usual dietary intake of lutein and zeaxanthin (L/Z).
   3. MPOD and serum L/Z concentration.
   4. Serum L/Z concentration and usual dietary intake of L/Z.
4. Multiple linear regression will be used to test for correlation to MPOD with the following variables:

   1. Daily hours of electronic device use.
   2. Usual dietary intake of L/Z.
   3. Age
   4. Gender

Results will be considered statistically significant if p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Male and females 18 to 65 years.
* Generally healthy.
* No participant reported history of clinically significant medical conditions including, but not limited to, cardiovascular, neurological, psychiatric, renal, immunological, endocrine (including uncontrolled diabetes or thyroid disease) or haematological abnormalities that are uncontrolled.
* Non-smoker

Exclusion Criteria:

* Participant reported diagnosis of serious ocular conditions (e.g. cataracts, glaucoma, diabetic retinopathy, retinitis pigmentosa, Stagardt's disease)
* Participant reported diagnosis, or current treatment of age-related macular degeneration.
* Participant reported diagnosis of epilepsy.
* Current or past smoker (within last 12 months).
* Under 18 or over 65 years of age.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy males and females, 18-65 years of age from Brisbane and surroudning areas, Australia.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Macular Pigment Optical Density | Triplicate measurement day 1
  Machine: Macular Pigment Screener II (Elektron Eye Technology). The non-invasive test uses heterochromatic flicker photometry.

SECONDARY OUTCOMES:
Dietary intake of lutein and zeaxanthin | Retrospective intake prior one month
  Daily intake of lutein and zeaxanthin (mg/day) measured by food frequency questionnaire.
Usual use of electronic devices. | Retrospective use of devices prior 3 months.
  Capturing exposure to blue light from electronic devices through questionnaire that asks participants to record usual hours of device use each day over last 3 months.
Blood lutein and zeaxanthin concentration | Single sample drawn on day of study visit (Day 1).
  Single sample of plasma to measure concentration of lutein and zeaxanthin by high performance liquid chromatography and photodiode array detection.

OTHER OUTCOMES:
Dietary intake of lutein and zeaxanthin on day prior to study visit. | Intake over single day prior to study visit (Day 1).
  24-hour diet recall to calculate dietary intake (mg/day) of lutein and zeaxanthin.

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Chachay, PhD, Principal Investigator — The University of Queensland
Locations (1):
- School of Human Movement and Nutrition Sciences, The University of Queensland, Saint Lucia, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chiu CJ, Chang ML, Zhang FF, Li T, Gensler G, Schleicher M, Taylor A. The relationship of major American dietary patterns to age-related macular degeneration. Am J Ophthalmol. 2014 Jul;158(1):118-127.e1. doi: 10.1016/j.ajo.2014.04.016. Epub 2014 Apr 29. PMID 24792100
- [Background] Wu J, Seregard S, Algvere PV. Photochemical damage of the retina. Surv Ophthalmol. 2006 Sep-Oct;51(5):461-81. doi: 10.1016/j.survophthal.2006.06.009. PMID 16950247
- [Background] Algvere PV, Marshall J, Seregard S. Age-related maculopathy and the impact of blue light hazard. Acta Ophthalmol Scand. 2006 Feb;84(1):4-15. doi: 10.1111/j.1600-0420.2005.00627.x. PMID 16445433
- [Background] Widomska J, Subczynski WK. Why has Nature Chosen Lutein and Zeaxanthin to Protect the Retina? J Clin Exp Ophthalmol. 2014 Feb 21;5(1):326. doi: 10.4172/2155-9570.1000326. PMID 24883226
- [Background] Stringham JM, Stringham NT, O'Brien KJ. Macular Carotenoid Supplementation Improves Visual Performance, Sleep Quality, and Adverse Physical Symptoms in Those with High Screen Time Exposure. Foods. 2017 Jun 29;6(7):47. doi: 10.3390/foods6070047. PMID 28661438
- [Background] Williams R, Bakshi S, Ostrin EJ, Ostrin LA. Continuous Objective Assessment of Near Work. Sci Rep. 2019 May 6;9(1):6901. doi: 10.1038/s41598-019-43408-y. PMID 31061427
- [Background] van der Veen RL, Berendschot TT, Hendrikse F, Carden D, Makridaki M, Murray IJ. A new desktop instrument for measuring macular pigment optical density based on a novel technique for setting flicker thresholds. Ophthalmic Physiol Opt. 2009 Mar;29(2):127-37. doi: 10.1111/j.1475-1313.2008.00618.x. PMID 19236582
- See also: Recruitment page with introductory information about study. — https://habs.uq.edu.au/research/volunteer-research-study/understanding-link-between-diet-chronic-device-light-exposure-and-eye-pigment